CLINICAL TRIAL: NCT03029546
Title: The Effect of Acute Glucose Loading on Level of Expression of Advanced Glycation End Products in Women Screened for Gestational Diabetes During Pregnancy
Brief Title: Effect of Glucose Load on Expression of Advanced Glycation End Products in Women Screened for Gestational Diabetes
Status: Completed | Type: Observational
Sponsor: Ohio State University (Other)
Collaborators: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Catalin S Buhimschi, MD, Principle Investigator, Ohio State University
Other Study IDs: 2015H0236
Record Dates: First submitted 2017-01-12; First posted 2017-01-24 (Estimated); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Inflammation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Glucose load: 50 subjects undergoing routine gestational diabetes screen with 50g glucose load.
  5 subjects undergoing follow-up gestational diabetes screen with 100g glucose load.
- Control: 50 subjects undergoing water ingestion with the same study measurements as the glucose load group at the same time intervals.

SUMMARY:
The investigator's main objective is to analyze the effects of a routine prenatal care screening tool (glucola test for gestational diabetes) on maternal inflammation through assessment of maternal circulatory biomarkers and blood pressure. Improving knowledge about routine prenatal care and how a variety of screening factors affect maternal physiology allows the investigators to be educated and informed when caring for mothers with medical co-morbidities.

* Determine if an acute glucose load (50g) is associated with an in-vivo and in-vitro increase in the concentration of Advanced Glycation End Products (AGEP's) that, in turn, can impact vascular endothelial reactivity and induce an acute increase in blood pressure. Previous studies generated in the investigators' laboratory showed that circulating soluble Receptor for Advanced Glycation End Products (sRAGE) and Tumor Necrosis Factor (TNF)-a (mediator of acute inflammation) are considered markers of the extent of maternal RAGE activation and/or systemic inflammation, respectively.
* Determine how an acute glucose load (50g) at the time of normal screening for gestational diabetes induces an acute increase in the level of sRAGE and TNF-a. If the investigators' hypothesis is confirmed, the investigators will have strong confirmation of the involvement of glycation products and TNF-a in generating the acute negative clinical symptoms of women experiencing a glucose tolerance test, such as headache, nausea, sweating, and bloating.

DETAILED DESCRIPTION:
A. Research Design Participants will be identified at the time of their prenatal care visit (24-28 weeks GA). The investigators will ask permission for participation in the research protocol. A waiver of HIPPA has been added to the protocol to explain the sources investigators might use to screen for eligible subjects. The electronic medical records may be accessed with a partial waiver to review the medical information that will make each subject a candidate for the protocol. The subject will be instructed on the benefits of the study for which the participant is eligible and that management will not be influenced by the participant's decision to volunteer or not. If the patient agrees to participate, the participant will be given the written consent to read. The participant will be asked if there is understanding, if all has been explained, and if there are any questions the investigators need to clarify. The informed consent will be obtained. No ads, flyers, website postings, recruitment letters, or oral/written scripts will be involved for recruitment of patients.

Interventions:

1. Informed consent.
2. Collection of blood (5 cc or one teaspoon of whole blood) and urine (1/2 cup) specimens prior to administration of the 50 gr. glucola test. This protocol will be presented in this arm of the study to women (n=50) who have a clinically indicated 1 hour glucose tolerance test to diagnose gestational diabetes.
3. Blood pressure measurements every 15 minutes for one hour.
4. Collection of a second blood (5 cc or one teaspoon of whole blood), and urine (1/2 cup) specimen following administration of the 50 gr. glucola test. Collection of blood at this time will be clinically indicated to test for abnormal clinical values that might classify the patient as gestational diabetic.
5. In a separate group of women classified as healthy pregnant controls (n=50) the investigators will obtain informed consent using a protocol similar to the one described above.
6. Collection of a blood (5 cc or one teaspoon of whole blood), and urine (1/2 cup) specimen will be performed prior to administration of the 50 cc of plain water.
7. Blood pressure measurements will be performed every 15 minutes for one hour.

d. Collection of a second blood (5 cc or one teaspoon of whole blood), and urine (1/2 cup) sample will occur at the end of the hour.

B. Sample Participants will be enrolled based on the eligibility for a one hour GTT. Chart reviews of the clinic schedules will be performed the week prior to identify the target population for recruitment who are 24-28 weeks gestation in need of a diabetes screen.

50 pregnant women in the high risk clinic presenting for diabetes screen at a routine prenatal visit will be recruited for enrollment. This population is at risk for subsequent adverse pregnancy outcomes, and the investigators will evaluate if biomarkers, such as advanced glycation end products, are affected following glucose loading for diabetes screening.

50 healthy pregnant women in the general obstetric clinic at McCampbell Hall will be recruited as controls to ingest a 50cc sample of water and undergo identical objective measurements (blood pressure measurements and urine/ blood samples) as the glucose loading subjects. Biomarker analysis will be compared with that of the glucose loading population. These patients serving as controls will undergo the clinically indicated glucola screening at another visit between 24-28 weeks gestation.

Exclusion criteria include:

1. Non-English-speaking subjects will be excluded due to inability to appropriately consent.
2. Non-pregnant patients will be excluded since this is a study of maternal tissues and pregnancy outcomes related to exposures in pregnancy.
3. Men will be excluded since this is a study that includes pregnant women only by nature of the research.
4. Prisoners will be excluded to avoid any potential for coercion
5. Minors under 18 years of age will be excluded due to lack of ability to consent without a legal guardian.
6. Patients with contra-indications to glucola testing for gestational diabetes screening will be excluded, such as bariatric surgery, inflammatory bowel disease with partial bowel resection, and other mal-absorptive conditions.

C. Measurement/ Instrumentation 50 pregnant patients who are 24 to 28 weeks gestation undergoing routine screening for gestational diabetes using a 50g glucose load will be recruited. Following enrollment, maternal blood and urine specimens will be obtained as outlined above. Blood pressure will be recorded. For this type of study design each patient will serve as the participant's own control. Additionally, 50 healthy pregnant patients will be recruited to perform a test similar to the diabetes screen using water only to serve as additional controls. Advanced Glycation End Products among other proteins will be analyzed for each of the specimens.

Using standard immunoassay procedures available in our laboratory, the investigators will perform in parallel proteomics analysis of urine and maternal blood in addition to placental evaluation following delivery. Advanced Glycation End Products and TNF-A will be the focus, but, by performing proteomics studies of the biological samples, the investigators hope to discover other biomarkers and biological pathways that might be responsible for the clinical manifestations of the test. The newly discovered key proteins and important regulatory protein pathways can potentially be targeted to identify and treat diabetes and other medical conditions in pregnancy.

D. Detailed Study Procedures Women will be recruited in the OSUMC High Risk or Low risk Clinics, and Labor and Delivery. Clinical data for the study will be abstracted from the subject's medical record.

Potential hazards are related to the risks of an additional blood draw outside of routine prenatal care. These risks include bruising, discomfort or pain at the site, infection, or fainting. The risks are perceived as minimal, but patients will be compensated for their time and willingness to undergo the discomfort of this additional blood draw.

Subjects will be coded as numbers 1 to 100. In addition, specimens will be coded with a letter code followed by numbers in consecutive number. The PI will create a computer worksheet where the name and medical record of the subject is linked to the coded information of the subject and to each of the coded specimen numbers. The computer desktop that holds the worksheet with Public Health Information (PHI) has a disk encryption. One copy of the consent form will be kept in a secured and locked cabinet in the PI's office which is also locked. The subject's name will be kept separate from the results. No reports will be communicated back to the subjects or included in their medical record, since they will not affect how pregnancy, labor or their post-delivery care will be managed. Only the subject's doctor and the researchers will know of the subject's participation in the study. No further public disclosure of this information will be made.

E. Internal Validity

To avoid study bias, we have also employed the following:

1. Use of internal controls and an external control group
2. Use of consecutive enrolled patients

F. Data Analysis Statistical comparisons between groups will be performed using Student t or Mann-Whitney test or Two-way repeated analysis of variance (ANOVA) followed by post hoc Holm-Sidak tests as appropriate. Pearson product moment correlation will be used to estimate association between variables. A p=<0.05 will be considered to indicate statistical significance. Gestational age, weight of the fetus at the time of glucose tolerance test, presence or absence of any of the medical complications of pregnancy, medication and substance abuse history, and maternal demographic characteristics will be analyzed and the subject of statistical comparison.

ELIGIBILITY:
Inclusion Criteria:

1. 50 pregnant women in the high risk clinic presenting for diabetes screen with 50g glucose load at a routine prenatal visit will be recruited for enrollment.
2. 5 pregnant women presenting for follow-up diabetes screen with 100g glucose load.

2. 50 healthy pregnant women in the general obstetric clinic at McCampbell Hall will be recruited as controls to ingest a 50cc sample of water and undergo identical objective measurements (blood pressure measurements and urine/ blood samples) as the glucose loading subjects.

Exclusion Criteria:

1. Non-English-speaking subjects will be excluded due to inability to appropriately consent.
2. Non-pregnant patients will be excluded since this is a study of maternal tissues and pregnancy outcomes related to exposures in pregnancy.
3. Men will be excluded since this is a study that includes pregnant women only by nature of the research.
4. Prisoners will be excluded to avoid any potential for coercion
5. Minors under 18 years of age will be excluded due to lack of ability to consent without a legal guardian.
6. Patients with contra-indications to glucola testing for gestational diabetes screening will be excluded, such as bariatric surgery, inflammatory bowel disease with partial bowel resection, and other mal-absorptive conditions.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women in the 2nd trimester eligible for gestational diabetes screening.
Sampling Method: Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
Concentration of advanced glycation end products in maternal serum following the glucose load | 1 hour following glucose load
  biomarker

CONTACTS AND LOCATIONS:
Overall Officials: Catalin Buhsimchi, MD, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jones ML, Buhimschi IA, Zhao G, Bartholomew A, Smith-Timms J, Rood KM, Buhimschi CS. Acute Glucose Load, Inflammation, Oxidative Stress, Nonenzymatic Glycation, and Screening for Gestational Diabetes. Reprod Sci. 2020 Aug;27(8):1587-1594. doi: 10.1007/s43032-020-00188-5. PMID 32430709
- [Derived] Jones ML, Buhimschi IA, Zhao G, Bartholomew A, Smith-Timms J, Rood KM, Buhimschi CS. Acute Glucose Load, Inflammation, Oxidative Stress, Nonenzymatic Glycation, and Screening for Gestational Diabetes. Reprod Sci. 2019 Feb 27:1933719119831772. doi: 10.1177/1933719119831772. Online ahead of print. PMID 30813845